CLINICAL TRIAL: NCT02463383
Title: Alcohol-related Breast Cancer in Postmenopausal Women - Effect of PPARG2pro12ala Polymorphism on Female Sex-hormone Levels and Interaction With Alcohol Consumption and NSAID Usage
Brief Title: Effect of PPARγ2 Polymorphism and NSAIDs on Acute Alcohol-induced Changes in Serum Estrogens Among Post-menopausal Women
Acronym: EPPNASE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Professor Lars Ove Dragsted (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Sponsor-Investigator, Professor Lars Ove Dragsted, Professor, Head of Section, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: M215
Record Dates: First submitted 2015-05-17; First posted 2015-06-04 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
Keywords: PPAR-gamma; estrogens; NSAIDS; polymorphism; metabolomics
MeSH Terms: conditions — Breast Neoplasms | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: Participants are randomized to an ibuprofen or placebo pill in the first period and are then provided with placebo or ibuprofen pills, respectively, in the second period in a crossover fashion. Alcohol (0.4g/kg bw) is provided as a challenge 30min after the pill has been swallowed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): 1. Ibuprofen Tab 400MG
  2. Placebo Tab
  Interventions: Drug: Ibuprofen Tab 400 MG; Drug: Placebo tab
- Sequence 2 (Experimental): 1. Placebo tab
  2. Ibuprofen Tab 400MG
  Interventions: Drug: Ibuprofen Tab 400 MG; Drug: Placebo tab

INTERVENTIONS:
Drug: Ibuprofen Tab 400 MG — 400mg ibuprofen is provided and an alcohol challenge (0.4g/kg bw) is given 30min later
  Other Names: (RS)-2-(4-(2-methylpropyl)phenyl)propanoic acid
Drug: Placebo tab — A placebo tablet is provided and an alcohol challenge (0.4g/kg bw) is given 30min later
  Other Names: placebo tablet

SUMMARY:
Postmenopausal women, stratified by a peroxisome proliferator-activated receptor gamma-2 (PPARG) polymorphism, were given the following treatments in a random order with a 5w wash-out period: a 400mg ibuprofen tablet or a placebo tablet; both treatments were followed after 30min by a single acute dose of 0.4g alcohol per kg bw. Serum estrogen levels were measured before and at three timepoints after alcohol intake. It is hypothesized that the acute decrease in estrogen sulphate and other markers of estrogens after alcohol intake is modulated by ibuprofen and by PPARG genotype.

DETAILED DESCRIPTION:
In a pilot human intervention trial we aimed to determine the effect of the PPARG Pro12Ala polymorphism and the PPARγ stimulator, Ibuprofen, on sex-hormone levels following alcohol intake in postmenopausal women. Seven women with PPARG Pro12Ala and 18 PPARG wildtype women were included.The study was performed as a randomised, double-blinded, placebo controlled 2x24 h crossover study. The volunteers were randomised to 1 of 2 groups who got the two treatments in different orders. Treatment 1 was a placebo tablet with water followed after 30min by an alcoholic drink providing 0,4g alcohol per kilogram bw and treatment 2 was an Ibuprofen tablet (400mg) with water followed by the same alcoholic drink. The two treatments were separated by a 5-7 weeks washout period. Alcohol was supplied as 7.7% ethanol in a lime-flavoured drink and was consumed over 15 min. EDTA-plasma was collected 40min before and 30, 60 and 90 min after ethanol intake as well as after 24 hours. Ibuprofen (400mg) was provided together with 100mL water 30min before the ethanol. Urine was collected throughout the 24 hour interval. Serum estrone, estrone sulphate, serum estrogen-binding globulin (SHBG), and ethanol were determined. It is hypothesized that the acute decrease in estrogen sulphate and other markers of estrogens after alcohol intake is modulated by ibuprofen and by PPARG genotype.

ELIGIBILITY:
Inclusion Criteria:

1. postmenopausal (last menses at least 1 year earlier);
2. having a weekly alcohol use of less than 14 drinks
3. having a BMI of 18-35;

Exclusion Criteria:

1. a history of alcohol abuse
2. alcohol abstaining
3. history of hysterectomy before last menses with preservation of both ovaries (unless a medical confirmation for the postmenopausal status exists or the participant is 60 years or older);
4. major health problems, such as ulcers, heart diseases, diabetes or cancer
5. previous or current use of HRT
6. taking prescription medications that could interfere with the study (i.e. daily use of NSAIDs and/or medication that interact with PPARγ e.g. cholesterol lowering medicine);
7. being allergic to alcohol and/or Ibuprofen
8. smoking

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Serum estrone sulphate (pmol/l) | from 40 min before to 90 min after alcohol consumption
  Plasma estrone sulfate concentration after acute ethanol intake by Ibuprofen intake and/or PPARG genotype

SECONDARY OUTCOMES:
Serum estrone (pmol/l) | from 40 min before to 90 min after alcohol consumption
  Plasma estrone decrease after acute ethanol intake by ibuprofen intake and/or PPARG genotype
Serum SHBG (nmol/l) | from 40 min before to 90 min after alcohol consumption
  Plasma SHBG concentration after acute ethanol ingestion by ibuprofen intake and/or PPARG genotype
Serum ethanol (g/l) | from 40 min before to 90 min after alcohol consumption
  Plasma ethanol concentration after acute ethanol ingestion
Serum metabolomics (relative metabolite intensity) | from 40 min before to 24h after alcohol intake
  The plasma metabolome profile by time after alcohol intake
Urine metabolomics (relative metabolite intensity) | from 40 min before to 24h after alcohol intake
  The urine metabolome profile by time after alcohol intake

CONTACTS AND LOCATIONS:
Overall Officials: Lars O Dragsted, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Derived] Kopp TI, Jensen DM, Ravn-Haren G, Cohen A, Sommer HM, Dragsted LO, Tjonneland A, Hougaard DM, Vogel U. Alcohol-related breast cancer in postmenopausal women - effect of CYP19A1, PPARG and PPARGC1A polymorphisms on female sex-hormone levels and interaction with alcohol consumption and NSAID usage in a nested case-control study and a randomised controlled trial. BMC Cancer. 2016 Apr 21;16:283. doi: 10.1186/s12885-016-2317-y. PMID 27102200